CLINICAL TRIAL: NCT00098280
Title: A Hemoglobin Stabilization and Transfusion Reduction Efficacy and Safety Clinical Investigation, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Using Eculizumab in Paroxysmal Nocturnal Hemoglobinuria Patients
Brief Title: Eculizumab to Treat Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050048; 05-H-0048
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-02

CONDITIONS: Hemoglobinuria, Paroxysmal
Keywords: H5g1; PNH; TRIUMPH; Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

INTERVENTIONS:
Drug: Eculizumab

SUMMARY:
This study will examine the safety and effectiveness of the experimental drug eculizumab in treating patients with paroxysmal nocturnal hemoglobinuria (PNH), a rare disorder of red blood cells that leads to premature destruction of the cells and resulting anemia. Patients may be at high risk of blood clots and may develop bone marrow failure or aplastic anemia, with low white blood cell and platelet counts. Eculizumab is a monoclonal antibody that may help improve the survival of red blood cells.

Patients 18 years of age and older with PNH who require blood transfusions for anemia and have received at least four transfusions in the 12 months preceding evaluation for this study may be eligible to enroll. Candidates are screened with a medical history, physical examination, and check of vital signs.

Participants have an electrocardiogram (EKG) and blood and urine tests, and are vaccinated against Neisseria meningitides, a common bacteria that can cause a disabling or fatal type of meningitis. They then enter an observation phase of the study, with monthly visits during which they complete a questionnaire; update their health status, transfusion record, and medication use; have their vital signs checked and PNH symptoms evaluated; have blood and urine tests; and receive a transfusion, if necessary. These visits continue for up to 3 months until patients receive a "qualifying" transfusion; that is, a transfusion given as a consequence of a certain hemoglobin level with symptoms or a different level without symptoms.

Patients are then randomly assigned to receive either eculizumab or a placebo (salt solution with no active ingredient). Both study medications are given intravenously (through a vein) over 30 minutes once a week for five doses and then once every 2 weeks for another 11 doses. At each treatment visit (study weeks 0-24), patients update their health status, transfusion records, and medication use; have their vital signs checked; and provide a blood sample. At various visits, they also complete a questionnaire, provide a urine sample and have an EKG. At the last treatment visit (week 26 or the final visit for patients who end their participation before visit 18) patients have a complete physical examination in addition to the procedures listed above.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is an acquired clonal disorder of the hematopoietic stem cell characterized by intravascular hemolysis, hemoglobinuria, anemia, and thrombosis. The clinical features of PNH result from the lack of one or more of the GPI-linked proteins that serve to protect cells from autologous complement mediated attack. Two such proteins, CD55 (decay accelerating factor) and CD59 (reactive lysis inhibitor) have been shown to be absent from PNH erythrocytes and platelets as well as other cell types.

Evidence strongly suggests that lack of the terminal complement inhibitor CD59 is responsible for the sensitivity of PNH erythrocytes and platelets to the effects of autologous complement. Since the pathogenesis of PNH is due to the inability of PNH red cells and platelets to inhibit the activation of terminal complement, it is logical to hypothesize that a terminal complement inhibitor could effectively stop the intravascular hemolysis, obviate or lessen the need for transfusions, and possibly decrease the propensity of life threatening thrombosis. Eculizumab is a humanized monoclonal antibody that like CD59 inhibits terminal complement.

This study is a randomized, double-blind, placebo controlled, multi-center study of eculizumab or placebo administered intravenously to approximately 75 PNH patients. The study is designed to evaluate the safety of eculizumab in transfusion dependent patients with paroxysmal nocturnal hemoglobinuria (PNH) and to determine if the administration of this terminal complement inhibitor could provide a safe and effective substitute for CD59 function.

ELIGIBILITY:
INCLUSION CRITERIA - Screening Period:

Individuals at least 18 years of age;

Patients must have required at least 4 episodes of transfusions in the 12 months prior to Visit 1 for anemia or anemia-related symptoms;

Presence of a GPI deficient red blood cell clone (type II cells) by flow cytometry of greater than or equal to 10%;

Patients taking erythropoietin must be on a stable dose for 26 weeks prior to visit 1 and the dose must be expected to remain stable during the Observation Period and the Treatment Phase;

Patients taking immunosuppressants must be on a stable dose for at least 26 weeks prior to Visit 1 and the dose must be expected to remain stable during the Observation period and the Treatment Phase;

Patients taking corticosteroids must be on a stable dose for at least 4 weeks prior to Visit 1. The dose level may be decreased during the study as clinically appropriate. If the corticosteroids need to be increased, they may not be increased above the dose reported at Visit 1;

Patients are allowed to take coumadin, but must be at a stable international normalized ratio (INR) level for 4 weeks prior to Visit 1 and are expected to maintain a stable INR level during the Observation Period and the Treatment Phase;

Patients taking iron supplements or folic acid must be on a stable dose for 4 weeks prior to Visit 3 and be expected to remain stable during Observation Period and the Treatment Phase;

Patients are allowed to take low molecular weight heparin, but must be on a stable dose for 4 weeks prior to Visit 1 and the dose must be expected to remain stable during Observation period and the Treatment Phase;

Patient must be willing and able to give written informed consent;

Patients must be vaccinated against N. meningitidis at Visit 1 or at least 14 days prior to Visit 3;

Patient must avoid conception during the trial using a method that is most appropriate for their physical state and culture.

INCLUSION CRITERIA - Observation Period:

Documented LDH level greater than or equal to 1.5 x upper limit of normal (ULN) either at Visit 1 or during the Observation Period;

Patients who have received one PRBC transfusion during the Observation Period at a hemoglobin value of less than or equal to 9 gm/dL with symptoms or at a hemoglobin value of less than or equal to 7 gm/dL without symptoms, and also within 1.5 gm/dL of the mean hemoglobin pre-transfusion value for the previous 12 months. This transfusion should be in accordance with that patient's individual transfusion hemoglobin algorithm, and occur within 48 hours of the hemoglobin sample that precipitated the transfusion;

Platelet count greater than or equal to 100,000/mm(3) either at Visit 1 or during the Observation Period.

EXCLUSION CRITERIA:

Patients whose mean hemoglobin levels prior to transfusion over the previous 12 months is greater than 10.5 gm/dL;

Absolute Neutrophil count less than or equal to 500/microL;

Presence or suspicion of active bacterial infection, in the opinion of the Investigator, at Visit 3 or recurrent bacterial infections;

Known or suspected hereditary complement deficiency;

Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days prior to Visit 1;

Pregnant, breast-feeding, or intending to conceive during the course of the study, including the Post-treatment Phase;

History of meningococcal disease;

History of bone marrow transplantation;

Any condition that, in the opinion of the Investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2004-12; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hillmen P, Lewis SM, Bessler M, Luzzatto L, Dacie JV. Natural history of paroxysmal nocturnal hemoglobinuria. N Engl J Med. 1995 Nov 9;333(19):1253-8. doi: 10.1056/NEJM199511093331904. PMID 7566002
- [Background] Tabbara IA. Hemolytic anemias. Diagnosis and management. Med Clin North Am. 1992 May;76(3):649-68. doi: 10.1016/s0025-7125(16)30345-5. PMID 1578962
- [Background] Rosse WF. Phosphatidylinositol-linked proteins and paroxysmal nocturnal hemoglobinuria. Blood. 1990 Apr 15;75(8):1595-601. No abstract available. PMID 2183885